CLINICAL TRIAL: NCT04359875
Title: Does a Systematic Phone-call by a Medical Student/General Practitioner Team in Patients Suffering From a Chronic Condition During the COVID-19 Containment Period Impact One-month Hospitalization's Rate in France? A Cluster Randomized Trial
Brief Title: A Phone-call With a Student/General Practitioner Team to Impact Morbidity of Chronic Patients During COVID-19 Containment
Acronym: COVIQuest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: INSERM CIC-P 1415 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-CD-COVIQuest (COVID-19); 2020-A01061-38 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-04-18; First posted 2020-04-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Diseases; Mental Disorder
Keywords: general practice; COVID-19; chronic diseases; medical student
MeSH Terms: conditions — Cardiovascular Diseases; Mental Disorders; COVID-19; Chronic Disease

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial with 2 subtrials : COVIQuest_CV and COVIQuest_MH.
  COVIQuest_CV involves patients ≥ 70 years old suffering from chronic cardiovascular disease; and COVIQuest_MH involves patients suffering from a mental health disease.
  As a note, both sub-trials are two-parallel group cluster randomized trials. Clusters will be defined as practices. Practices will be randomized into two groups A and B. For practices in group A: their CV patients constitute the experimental group for the COVIQuest_CV trial, their MH patients constitute the control group for the COVIQuest_MH trial. For practices in group B: their CV patients constitute the control group for the COVIQuest_CV trial, their MH patients constitute the experimental group for the COVIQuest_MH trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Management by a student/general practitioner tandem (Experimental): Patients will receive a phone call from the medical student who will inquire about their health. The medical student will then transmit this information to the general practitioner who will decide on the most suitable management for the patient.
  Interventions: Behavioral: Phone-call screening and management by a medical student/general practitioner tandem
- Usual care (No Intervention): Usual care, i.e. patients will call their general practitioner when needed, up to 1 month, which corresponds to the estimated time for the intervention to be delivered to all patients in the intervention group.
  At the end of the intervention at 1 month, patients in the usual care group will also receive a phone-call from the medical student/general practitioner tandem.

INTERVENTIONS:
Behavioral: Phone-call screening and management by a medical student/general practitioner tandem — Systematic phone contact of the patient by a medical student, under the indirect supervision of the general practitioner. This phone contact will be standardized with 3 questions to ask to the patient:
  * How are you doing? (with a Likert scale from 1=very bad to 10=very well)
  * Would you have made an appointment with your general practitioner if there had not been COVID19 epidemic and containment?
  * Would you like an appointment with your doctor and / or has your doctor ever contacted you? In view of the answers to these 3 questions, the general practitioner will decide whether it is necessary to propose a consultation or a teleconsultation to the patient, taking into account his/her medical background.
  Arms: Management by a student/general practitioner tandem

SUMMARY:
Following the announcement of the containment of the population due to the COVID-19 epidemic on March 17, 2020 in France, a notable decrease in the number of consultations in general practice was reported. Patients no longer contact their general practitioner, including those with regular follow-up for one or more chronic conditions. This observation raised worries since it could lead to delay or failure in detecting decompensations / complications of these chronic conditions by a lack of recourse to care. Thus, an urgent message from the National Health Department (Direction Générale de la Santé - DGS) was adressed on April 8, 2020 to the health professionals regarding the organization of care aside from COVID-19. The main recommendation was "that the personal physician or the corresponding specialist should contact the most fragile patients with chronic condition to ensure follow-up and detect any risk of decompensation ".

Such fragile patients are in great numbers, up to more than 200 for an average general practitioner. Therefore, although this recommendation is regarded as "essential in view of the health needs of the population", it will prove quite difficult to follow without the help of a skilled external assistance that can be quickly mobilized.

DETAILED DESCRIPTION:
Following the announcement of the containment of the population due to the COVID-19 epidemic on March 17, 2020 in France, a notable decrease in the number of consultations in general practice was reported. Patients no longer contact their general practitioner, including those with regular follow-up for one or more chronic conditions. This observation raised worries since it could lead to delay or failure in detecting decompensations / complications of these chronic conditions by a lack of recourse to care. Thus, an urgent message from the National Health Department (Direction Générale de la Santé - DGS) was adressed on April 8, 2020 to the health professionals regarding the organization of care aside from COVID-19. The main recommendation was "that the personal physician or the corresponding specialist should contact the most fragile patients with chronic condition to ensure follow-up and detect any risk of decompensation ".

Such fragile patients are in great numbers, up to more than 200 for an average general practitioner. Therefore, although this recommendation is regarded as "essential in view of the health needs of the population", it will prove quite difficult to follow without the help of a skilled external assistance that can be quickly mobilized.

The COVIQUEST project is a cluster randomized trial in general practice designed to assess the optimizationg of the screening and management of patients with chronic condition at risk of decompensation through a collaboration between the general practitioner and a medical student.

The trial will focus on patients wit cardiovascular conditions aged 70 or more and patients with mental health conditions. These conditions are both highly prevalent in general practice and both at risk of severe short-term complications.

Practices will be randomly assigned to a group (A or B). In group A, students will start by contacting patients with cardiovascular conditions; in group B they will start by contacting patients patients with mentral health conditions. The students will call these patients on the phone and ask them specific questions about their health, their needs, and if they want their general practitioner to call them back. The student will then transmit this information to the general practitioner who will decide on the best care to offer the patient.

The primary outcome is defined as the occurrence of hospitalization during a one-month period after the phone call. It will be collected by a second phone call from the medical student. This time, all patients will be contacted, i.e. both patients with mental illness and cardiovascular patients, whatever the group. Thus, patients allocated to the control groups (i.e. patients with mental illness from group A and cardiovascular patients from group B) will also benefit from the intervention at 1 month: again, students will ask patients about their health and whether they want their general practitioner to call them back.

This approach has several advantages:

1. all patients will benefit from a phone call, in accordance with the recommendations of the DGS,
2. the involvement of students, competent in medical interviews and quickly mobilizable, will help general practitioners, on the front line of many missions, without any health risk linked to the contagiousness of COVID-19 for students,
3. randomizing the call order will allow to assess with a high level of evidence the impact of such an organization on hospitalizations, for two families of diseases with high prevalence.

The trial will involve at least nine French regions. Considering that the general practitioner's patient base numbers an average of 110 patients with chronic cardiovascular disease or chronic mental illness, and that at least 25 general practitioners per region participate in the study, we can expect that 22,000 patients will benefit from the intervention of this study.

ELIGIBILITY:
Inclusion criteria (patient with a chronic cardiovascular) :

* Male or female
* >= 70 years of age
* Participants covered by or entitled to social security
* With a chronic cardiovascular or mental disease as referenced in the long term illness (ALD) list (i.e. with an ALD n°1, 3, 5, 12, 13 for cardiovascular disease)
* Followed regularly by their general practitioner (i.e. entered in the list of patients followed by a general practitioner by French Health Insurance
* Participants who has given oral, express and informed consent.

Inclusion criteria (patient with a mental disease) :

* Male or female
* >= 18 years of age
* Participants covered by or entitled to social security
* With a chronic cardiovascular or mental disease as referenced in the long term illness (ALD) list (i.e. with an ALD 23 for mental disease)
* Followed regularly by their general practitioner (i.e. entered in the list of patients followed by a general practitioner by French Health Insurance
* Participants who has given oral, express and informed consent

Exclusion criteria :

* Patients with both a cardiovascular ALD and a mental health ALD (they will benefit from the intervention, without participating in the trial)
* Patients already and directly managed by their general practitioner during containment and whose general practitioner refuses that the patient be contacted by someone other than himself
* Patients unable to provide informed consent.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22000 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Hospitalization(s) at 1 month | 1 month
  Hospitalization over a one month period. The primary outcome will be collected by a phone call from a medical student to the patient 1 month after randomization date. Hospitalizations (date, location, length, if available, and reason) will be collected. Because there will be many patients to be called for each practitioner, we expect these phone call to occur within a few days after day 28.

SECONDARY OUTCOMES:
Phone-call from the general practitioner (in the experimental group only) | 1 month
  In the experimental group only: proportion of patients for whom the practitioner had to call back after the medical student had phoned (just after allocation of the practice to the experimental group) at 1 month.
Mortality at 1 month | 1 month
  Mortality will be reported after checking with the city of the patient's home if there is no response to the phone call
Use of primary care | 6 months
  Number of general practitioner consultations and teleconsultations (and time of general practitioner consultation, i.e. during the containment period or not) using data from the French Health National (SNDS) Database
Use of secondary care | 6 months
  Number of consultations with another medical specialist (and time of consultation, i.e. during the containment period or not) using data from the French Health National (SNDS) Database
Number of prescriptions related to the chronic disease dispensed by the pharmacy | 6 months
  Number of prescriptions related to the chronic disease that were dispensed by the pharmacy using data from the French Health National (SNDS) Database
Number of hospitalization(s) | 6 months
  Number of hospitalizations using data from the French Health National (SNDS) Database
Time to hospitalization(s) | 6 months
  Time to hospitalization using data from the French Health National (SNDS) Database
Hospitalization(s)' durations | 6 months
  Hospitalization duration using data from the French Health National (SNDS) Database
Reasons for hospitalization(s) | 6 months
  Reason for hospitalization using data from the French Health National (SNDS) Database
Mortality at 6 months | 6 months
  Number of deaths using data from the French Health National (SNDS) Database
Cardiovascular events (MACE) | 6 months
  Only for patients in the COVIQuest_CV sub-trial: Cardiovascular events (MACE): nonfatal stroke, nonfatal myocardial infarction, cardiovascular death and hospitalization for heart failure using data from the French Health National (SNDS) Database
Psychotropic drugs | 6 months
  Only for patients in the COVIQuest_MH sub-trial: Psychotropic drugs consumption using data from the French Health National (SNDS) Database

CONTACTS AND LOCATIONS:
Overall Officials: CLARISSE DIBAO-DINA, MD-PhD, Study Director — University Hospital of TOURS
Locations (1):
- Dibao-Dina, Tours, France

IPD SHARING:
Plan to Share IPD: Yes
One-month-data can be shared, whereas 6-month data are not legally sharable (electronic health records).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: email

REFERENCES:
- [Result] Sauvage A, Laurent E, Giraudeau B, Tassi MF, Godillon L, Grammatico-Guillon L, Dibao-Dina C. Six-month outcomes after a GP phone call during the first French COVID-19 lockdown (COVIQuest): a cluster randomised trial using medico-administrative databases. BMJ Open. 2024 Nov 24;14(11):e085094. doi: 10.1136/bmjopen-2024-085094. PMID 39581719
- [Derived] Dibao-Dina C, Leger J, Ettori-Ajasse I, Boivin E, Chambe J, Abou-Mrad-Fricquegnon K, Sun S, Jego M, Motte B, Chiron B, Sidorkiewicz S, Khau CA, Bouchez T, Ghali M, Bruel S, Lebeau JP, Camus V, El-Hage W, Angoulvant D, Caille A, Guillon-Grammatico L, Laurent E, Saint-Lary O, Boussageon R, Pouchain D, Giraudeau B; COVIQuest group. Impact of a phone call with a medical student/general practitioner team on morbidity of chronic patients during the first French COVID-19 lockdown (COVIQuest): a cluster randomised trial. BMJ Open. 2022 Jul 28;12(7):e059464. doi: 10.1136/bmjopen-2021-059464. PMID 35902188